CLINICAL TRIAL: NCT03075163
Title: Optimization of Post-Operative Therapy for Nausea or Vomiting
Brief Title: Post-Operative Therapy for Nausea or Vomiting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment futility
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 932163
Record Dates: First submitted 2017-01-11; First posted 2017-03-09 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Vomiting; Nausea
Keywords: PONV; Nausea; Vomiting; Acupressure
MeSH Terms: conditions — Vomiting; Nausea; Postoperative Nausea and Vomiting | interventions — Acupressure; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental): Manual pressure will be applied on the wrists bilaterally.
  Interventions: Procedure: Acupressure
- Ondansetron (Active Comparator): Ondansetron (Zofran) is used for the treatment of nausea and vomiting.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Procedure: Acupressure — Specifically trained personnel will apply pressure on the wrists bilaterally at the P6 point for up to 3 minutes. The P6 point is located three fingerbreadths from the wrist crease on the volar surface of the arm between the palmaris longus and flexor carpi radialis.
  In the event of failure in the acupressure group, further treatments will be identical to the control group. Since Ondansetron is the standard Post Anesthetic Care Unit treatment, it will be first line rescue therapy except in the case that the patient has received 8mg in the past 6 hours. If needed, further antiemetic pharmacologic treatments may include, but are not limited to, phenergan, metoclopramide, haloperidol, diphenhydramine or propofol at the clinical discretion of the patient's anesthesiology care team.
  Arms: Acupressure
Drug: Ondansetron — Ondansetron is a medication that belongs to the drug class known as antiemetic and selective 5-HT3 receptor antagonist. Ondansetron is prescribed for the treatment of nausea and vomiting due to cancer chemotherapy and also used to prevent and treat nausea and vomiting after surgery.
  Other Names: Zofran
  Arms: Ondansetron

SUMMARY:
This is a single site, prospective, randomized controlled study designed to evaluate the impact of acupressure when used as an initial treatment before rescue medications in the treatment of post-operative nausea and/or vomiting at UCD.

DETAILED DESCRIPTION:
Each individual will only participate in the post anesthetic care unit starting from when the patient's nurse or anesthesiology team deems that the patient needs treatment for PONV. It ends when the patient is discharged from anesthesiology care.

Patients will be asked to score nausea before randomized treatment of acupressure or medication, and to score nausea after treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for elective surgery requiring general anesthesia

Exclusion Criteria:

* Age less than 18 years
* Adults unable to give primary consent
* Pregnancy
* Prisoners
* Unable to access pericardial 6 acupressure point bilaterally post procedure
* Allergy to Ondansetron

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Marc, MD, PhD, Principal Investigator — University of CA, Davis; Neal W Fleming, MD, PhD, Principal Investigator — University of CA, Davis
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parra-Sanchez I, Abdallah R, You J, Fu AZ, Grady M, Cummings K 3rd, Apfel C, Sessler DI. A time-motion economic analysis of postoperative nausea and vomiting in ambulatory surgery. Can J Anaesth. 2012 Apr;59(4):366-75. doi: 10.1007/s12630-011-9660-x. Epub 2012 Jan 6. PMID 22223185
- [Background] Chandrakantan A, Glass PS. Multimodal therapies for postoperative nausea and vomiting, and pain. Br J Anaesth. 2011 Dec;107 Suppl 1:i27-40. doi: 10.1093/bja/aer358. PMID 22156268
- [Background] Hirsch J. Impact of postoperative nausea and vomiting in the surgical setting. Anaesthesia. 1994 Jan;49 Suppl:30-3. doi: 10.1111/j.1365-2044.1994.tb03580.x. PMID 8129160
- [Background] Gan TJ, Meyer TA, Apfel CC, Chung F, Davis PJ, Habib AS, Hooper VD, Kovac AL, Kranke P, Myles P, Philip BK, Samsa G, Sessler DI, Temo J, Tramer MR, Vander Kolk C, Watcha M; Society for Ambulatory Anesthesia. Society for Ambulatory Anesthesia guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2007 Dec;105(6):1615-28, table of contents. doi: 10.1213/01.ane.0000295230.55439.f4. PMID 18042859
- [Background] White PF, Zhao M, Tang J, Wender RH, Yumul R, Sloninsky AV, Naruse R, Kariger R, Cunneen S. Use of a disposable acupressure device as part of a multimodal antiemetic strategy for reducing postoperative nausea and vomiting. Anesth Analg. 2012 Jul;115(1):31-7. doi: 10.1213/ANE.0b013e3182536f27. Epub 2012 Apr 13. PMID 22504214
- [Background] Lee A, Fan LT. Stimulation of the wrist acupuncture point P6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003281. doi: 10.1002/14651858.CD003281.pub3. PMID 19370583
- [Background] Liodden I, Howley M, Grimsgaard AS, Fonnebo VM, Borud EK, Alraek T, Norheim AJ. Perioperative acupuncture and postoperative acupressure can prevent postoperative vomiting following paediatric tonsillectomy or adenoidectomy: a pragmatic randomised controlled trial. Acupunct Med. 2011 Mar;29(1):9-15. doi: 10.1136/aim.2010.002915. Epub 2010 Dec 18. PMID 21169634
- [Background] Alessandrini M, Napolitano B, Micarelli A, de Padova A, Bruno E. P6 acupressure effectiveness on acute vertiginous patients: a double blind randomized study. J Altern Complement Med. 2012 Dec;18(12):1121-6. doi: 10.1089/acm.2011.0384. Epub 2012 Sep 5. PMID 22950829
- [Background] Noroozinia H, Mahoori A, Hasani E, Gerami-Fahim M, Sepehrvand N. The effect of acupressure on nausea and vomiting after cesarean section under spinal anesthesia. Acta Med Iran. 2013 Apr 6;51(3):163-7. PMID 23605600
- [Background] Genc F, Tan M. The effect of acupressure application on chemotherapy-induced nausea, vomiting, and anxiety in patients with breast cancer. Palliat Support Care. 2015 Apr;13(2):275-84. doi: 10.1017/S1478951514000248. Epub 2014 Apr 30. PMID 24787745
- [Background] Huang ST, Chen GY, Lo HM, Lin JG, Lee YS, Kuo CD. Increase in the vagal modulation by acupuncture at neiguan point in the healthy subjects. Am J Chin Med. 2005;33(1):157-64. doi: 10.1142/S0192415X0500276X. PMID 15844844
- [Background] Tokumaru O, Chen JD. Effects of acupressure on gastric myoelectrical activity in healthy humans. Scand J Gastroenterol. 2005 Mar;40(3):319-25. doi: 10.1080/00365520410009636. PMID 15934175
- See also: Ondansetron — https://medlineplus.gov/druginfo/meds/a601209.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupressure: Manual pressure will be applied on the wrists bilaterally.
  Acupressure: Specifically trained personnel will apply pressure on the wrists bilaterally at the P6 point for up to 3 minutes. The P6 point is located three fingerbreadths from the wrist crease on the volar surface of the arm between the palmaris longus and flexor carpi radialis.
  In the event of failure in the acupressure group, further treatments will be identical to the control group. Since Ondansetron is the standard Post Anesthetic Care Unit treatment, it will be first line rescue therapy except in the case that the patient has received 8mg in the past 6 hours. If needed, further antiemetic pharmacologic treatments may include, but are not limited to, phenergan, metoclopramide, haloperidol, diphenhydramine or propofol at the clinical discretion of the patient's anesthesiology care team.
Period: Overall Study
Arm/Group | Acupressure | Ondansetron
Started | 150 | 150
Completed | 12 | 12
Not Completed | 138 | 138
Not completed — not eligible for treatment limb | 138 | 138

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupressure | Ondansetron | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Nausea Score
Description: Difference in the nausea score before and after treatment. Nausea is scored on a scale from 1 to 10 with 1 being no nausea and 10 being severe nausea with impending vomiting.
  A greater difference is indicative of a better outcome
Time Frame: Time to discharge from post anesthetic care unit
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Acupressure | Ondansetron
Number analyzed (Participants) | 12 | 12
score on a scale | 1.88 (1.8) | 1.25 (2.5)

ADVERSE EVENTS:
Time Frame: Time from completion of the surgical procedure and arrival in the post anesthetic care unit until discharge from the post anesthesia care unit
Description: Data collected from chart review
Arm/Group | Acupressure | Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT03075163/Prot_000.pdf